CLINICAL TRIAL: NCT02386241
Title: Identification of Genomic Changes in Families Having Multiple Members With Tumors
Status: Terminated | Type: Observational
Why Stopped: PI departure without replacement
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Translational Genomics Research Institute (Other)
Responsible Party: Principal Investigator, Lori Wood, Research Operations Manager, St. Joseph's Hospital and Medical Center, Phoenix
Other Study IDs: 14BN108
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Glioma
Keywords: brain tumor
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A single saliva or blood sample measuring 10mL for genomic analysis.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: saliva or blood sample collection — Single saliva or blood sample measuring 10mL for genomic analysis.

SUMMARY:
This study will compare genomic alterations between the parents and the patients with high-grade glioma.

DETAILED DESCRIPTION:
Genomic changes leading to the formation of brain tumors are slowly being discovered. Despite advances in genomic technology, much analysis is hindered by the lack of control samples that could better delineate genomic alterations leading to disease. The ideal genomic control would be the genetic material of the parents of afflicted individuals. The researchers propose to then compare the genomic material from parents of siblings, both of whom have a diagnosis of a high-grade glioma. Additionally, the researchers will then compare the genomic alterations between the parents and the patients. This analysis will provide an unprecedented insight into genomic level changes that take place between parents and patients that resulted in the formation of a high-grade glioma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Family history of brain tumor in first degree relative

Exclusion Criteria:

* less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Families having multiple members (1st degree) with tumors.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2015-03; Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Total genomic sequencing | within 30 days of blood or saliva collection
  Researchers will perform total genomic sequencing using next generation sequencing technology to identify common variants associated with familial brain tumors. Upon sequencing of the genomic material, the data analysis will be done using standard statistical methods. We will use bioinformatics tools (high throughput sequencing of genome) to identify genomic changes between parents and patients.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nakaji, MD, Principal Investigator — Saint Joseph's Hospital and Medical Center/Barrow Neurological Institute
Locations (1):
- Barrow Neurological Institute at St. Joseph's Hospital Medical Center, Phoenix, Arizona, United States